CLINICAL TRIAL: NCT01761994
Title: The Effect of Nafamostat Mesilate in Prolonging Filter Patency With Patients on Continuous Renal Replacement Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2007-0220
Record Dates: First submitted 2012-12-24; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Acute Kidney Injury
Keywords: nafamostat mesilate; heparin; continuous renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury | interventions — nafamostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- M100 (Active Comparator): heparin free CRRT group
  Interventions: Drug: Anticoagulation with nafamostat mesilate
- HF1000 (Experimental): CRRT with nafamostat mesilate anticoagulation group
  Interventions: Drug: Anticoagulation with nafamostat mesilate

INTERVENTIONS:
Drug: Anticoagulation with nafamostat mesilate — Initial dose of nafamostat mesilate is 20mg/hr. Dosage is adjusted from 10mg to 30mg/hr according to patients' status. For priming, two vial of nafamostat mesilate was dissolved in 2mL of 5% glucose fluid, and then mixed with 1000mL of normal saline. After carefully removing air bubble from the circuit with the prepared fluid, nafamostat mesilate was dissolved with 15 mL of 5% glucose fluid and loaded in anticoagulation line with starting dose of 20mg/hr.
  Other Names: futhan

SUMMARY:
Continuous renal replacement therapy (CRRT) has been considered as an effective modality for renal replacement therapy in hemodynamically unstable patients within intensive care unit (ICU) except for the necessity of anticoagulation. The severity and peculiarities of ICU patients often make it equivocal to use anticoagulation. This is a prospective randomized controlled study to show the difference in filter life span and adverse event between HF1000 (nafamostat mesilate) group and M100 (heparin-free) group.

ELIGIBILITY:
Inclusion Criteria:

* patients who have at least one of the hemorrhagic tendencies of following conditions and needs CRRT hemodynamically;

  1. Platelet count < 100,000
  2. aPTT > 60 sec
  3. PT-INR > 2.0
  4. active hemorrhage
  5. surgery within 48 hours
  6. cerebral hemorrhage within 3 months or history of major bleeding
  7. septic shock or DIC.

Exclusion Criteria:

* pregnancy, breast feeding, possibility of pregnancy,
* allergy to nafamostat mesilate,
* other conditions that physician consider unfit for candidate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
mortality | 2 years
  Mortality in intensive care unit

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Tsujimoto H, Tsujimoto Y, Nakata Y, Fujii T, Takahashi S, Akazawa M, Kataoka Y. Pharmacological interventions for preventing clotting of extracorporeal circuits during continuous renal replacement therapy. Cochrane Database Syst Rev. 2020 Dec 14;12(12):CD012467. doi: 10.1002/14651858.CD012467.pub3. PMID 33314078
- [Derived] Lee YK, Lee HW, Choi KH, Kim BS. Ability of nafamostat mesilate to prolong filter patency during continuous renal replacement therapy in patients at high risk of bleeding: a randomized controlled study. PLoS One. 2014 Oct 10;9(10):e108737. doi: 10.1371/journal.pone.0108737. eCollection 2014. PMID 25302581